CLINICAL TRIAL: NCT05009056
Title: Post-surgical Stability in Mandibular Advancement Using Postsurgical Versus Presurgical Computer Guided Functional Appliance. (RANDOMIZED CLINICAL TRIAL)
Brief Title: Functional Appliance for Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mokhtar Elsayed Hafez, Assistant Lecturer of Oral and Maxillofacial Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orthognathic surgery
Record Dates: First submitted 2021-08-04; First posted 2021-08-17 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Orthognathic Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- postsurgical computer guided functional appliance (Experimental): After achieving ideal condylar poison by computer guided surgery. The distal extension of the final occlusal wafer will be cut and the appliance will be fitted to be utilized as a postsurgical functional appliance for condylar adaptation. Patients will be instructed to wear the splints continuously for 3 months, only being allowed to remove them when eating and brushing their teeth.
  Interventions: Device: Postsurgical computer guided functional appliance
- Presurgical computer guided functional appliance (Active Comparator): Using the software, 3D digitized mandible will be virtually repositioned in ideal centric relation through accurate adjustment of the condyle in its glenoid fossa. Patients' dental casts will be scanned, and digitized into a virtual 3D model and superimposed to the CT cuts into the virtual plan software environment in order to produce preoperative CAD/CAM splint on the adjusted centric occlusion. Patients will be instructed to wear the splints continuously for 3 months, only being allowed to remove them when eating and brushing their teeth.
  Interventions: Device: Postsurgical computer guided functional appliance

INTERVENTIONS:
Device: Postsurgical computer guided functional appliance — After achieving ideal condylar poison by computer guided surgery. The distal extension of the final occlusal wafer will be cut and the appliance will be fitted to be utilized as a postsurgical functional appliance for condylar adaptation. Patients will be instructed to wear the splints continuously for 3 months, only being allowed to remove them when eating and brushing their teeth.

SUMMARY:
The unstable condylar position in the glenoid fossa is a critical problem for postsurgical instability after mandibular advancement with subsequent mandibular relapse. The habitual forward occlusion in class II patients creates unstable condyle to glenoid fossa relationship making it hard for clinicians to determine the amount of mandibular advancement. Splint therapy is considered as a preoperative reversible nonsurgical condylar repositioning option in addition to its adjunctive effect for pain relief in TMJ symptomatic patients. To minimize this relapse, presurgical functional appliance therapy has been proposed and has shown promising outcomes.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of postsurgical versus presurgical computer guided functional appliance in relapse prevention after mandibular advancement surgery.

Surgical procedure:

1. Owbgeser incision will be performed to expose the buccal and lingual aspects of the ramus angle region.
2. CAD/CAM generated preoperative wafer will be placed on the lower arch dentition, the guide has an extension to guide medial, vertical, oblique cuts as well as screw holes for reference landmarks for proximal segment & tooth bearing segment.
3. Drilling of all the reference landmarks on the proximal segment and locating medial, vertical, oblique cuts.
4. Removal of guide, then BSSO is performed.
5. The final wafer is placed, the guiding hole on the proximal segment will then be realigned with the previously drilled screw holes, fixation using mono cortical screws then drilling screw holes for plate fixation.
6. Fixation of the osteotomy using 2.0 mm pre-bent mini plates.
7. A positioning screw will be added to improve stability against rotational forces.

b-Functional appliance

Postsurgical computer guided functional appliance:

After achieving ideal condylar poison by computer guided surgery. The distal extension of the final occlusal wafer will be cut and the appliance will be fitted to be utilized as a postsurgical functional appliance for condylar adaptation. Patients will be instructed to wear the splints continuously for 3 months, only being allowed to remove them when eating and brushing their teeth.

Presurgical computer guided functional appliance:

Using the software, 3D digitized mandible will be virtually repositioned in ideal centric relation through accurate adjustment of the condyle in its glenoid fossa. Patients' dental casts will be scanned, and digitized into a virtual 3D model and superimposed to the CT cuts into the virtual plan software environment in order to produce preoperative CAD/CAM splint on the adjusted centric occlusion. Patients will be instructed to wear the splints continuously for 3 months, only being allowed to remove them when eating and brushing their teeth.

c- Follow up

All patients will be advised to stay on a soft diet for 4-6 weeks to avoid any undue forces on the surgical site. Postoperative CT and lateral cephalogram will be obtained, immediately postoperative and 12 months later respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patient above 18 years
* Patients in need of bilateral sagittal split osteotomy for mandibular advancement.
* All patients are free from any systemic disease that may affect normal bone healing.
* Sufficient dentition to reproduce the occlusal relationships
* Patient's consent to participate

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing
* Intra-bony lesions or infections that may interfere with surgery
* Previous orthognathic surgeries

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change from postoperative sagital position of the mandible at 12 months (skeletal stability) | immediately postoperative and 12 months later
  Method of Measurement: Lateral cephalogram Unit of Measurement: mm

SECONDARY OUTCOMES:
Assessment of condylar deviation | immediately postoperative and 12 months later
  Method of Measurement: CT scan Unit of Measurement: mm

OTHER OUTCOMES:
Distal segment linear deviation | immediately postoperative and 12 months later
  Method of Measurement: CT scan Unit of Measurement: mm
Distal segment angular deviations | immediately postoperative and 12 months later
  Method of Measurement: CT scan Unit of Measurement: degree

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic of Oral and Maxillofacial Surgery department- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ha N, Hong Y, Qu L, Chung M, Qu R, Cai X, Fang B, Jiang L. Evaluation of post-surgical stability in skeletal class II patients with idiopathic condylar resorption treated with functional splint therapy. J Craniomaxillofac Surg. 2020 Mar;48(3):203-210. doi: 10.1016/j.jcms.2020.01.004. Epub 2020 Jan 11. PMID 32008874
- [Background] Bailey L', Cevidanes LH, Proffit WR. Stability and predictability of orthognathic surgery. Am J Orthod Dentofacial Orthop. 2004 Sep;126(3):273-7. doi: 10.1016/S0889540604005207. No abstract available. PMID 15356484
- [Background] Proffit WR, Turvey TA, Phillips C. The hierarchy of stability and predictability in orthognathic surgery with rigid fixation: an update and extension. Head Face Med. 2007 Apr 30;3:21. doi: 10.1186/1746-160X-3-21. PMID 17470277
- [Background] Costa F, Robiony M, Toro C, Sembronio S, Polini F, Politi M. Condylar positioning devices for orthognathic surgery: a literature review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Aug;106(2):179-90. doi: 10.1016/j.tripleo.2007.11.027. Epub 2008 Apr 16. PMID 18417381
- [Background] TRAUNER R, OBWEGESER H. The surgical correction of mandibular prognathism and retrognathia with consideration of genioplasty. II. Operating methods for microgenia and distoclusion. Oral Surg Oral Med Oral Pathol. 1957 Sep;10(9):899-909. doi: 10.1016/s0030-4220(57)80041-3. No abstract available. PMID 13465100
- [Background] Bell WH, Schendel SA. Biologic basis for modification of the sagittal ramus split operation. J Oral Surg. 1977 May;35(5):362-9. PMID 403263
- [Background] Wyatt WM. Sagittal ramus split osteotomy: literature review and suggested modification of technique. Br J Oral Maxillofac Surg. 1997 Apr;35(2):137-41. doi: 10.1016/s0266-4356(97)90691-4. PMID 9146874
- [Background] Joss CU, Vassalli IM. Stability after bilateral sagittal split osteotomy advancement surgery with rigid internal fixation: a systematic review. J Oral Maxillofac Surg. 2009 Feb;67(2):301-13. doi: 10.1016/j.joms.2008.06.060. PMID 19138603
- [Background] Epker BN, Wessberg GA. Mechanisms of early skeletal release following surgical advancement of the mandible. Br J Oral Surg. 1982 Sep;20(3):175-82. doi: 10.1016/s0007-117x(82)80035-8. PMID 6958313
- [Background] Worms FW, Speidel TM, Bevis RR, Waite DE. Posttreatment stability and esthetics of orthognathic surgery. Angle Orthod. 1980 Oct;50(4):251-73. doi: 10.1043/0003-3219(1980)0502.0.CO;2. PMID 6935978
- [Background] Angle AD, Rebellato J, Sheats RD. Transverse displacement of the proximal segment after bilateral sagittal split osteotomy advancement and its effect on relapse. J Oral Maxillofac Surg. 2007 Jan;65(1):50-9. doi: 10.1016/j.joms.2005.11.117. PMID 17174764
- [Background] Nebbe B, Brooks SL, Hatcher D, Hollender LG, Prasad NG, Major PW. Interobserver reliability in quantitative MRI assessment of temporomandibular joint disk status. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Dec;86(6):746-50. doi: 10.1016/s1079-2104(98)90215-3. PMID 9868736